CLINICAL TRIAL: NCT06492629
Title: Phase II Clinical Study of Toripalimab Combined With Chidamide for the Treatment of Relapsed/Refractory Peripheral T-Cell Lymphoma
Brief Title: Toripalimab Combined With Chidamide for the Treatment of Relapsed/Refractory Peripheral T-Cell Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, SHENGYANG, Director, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTCL-001
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: PTCL
MeSH Terms: interventions — toripalimab; N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Toripalimab Combined With Chidamide group (Experimental): Toripalimab:Intravenous infusion, 240mg, administered once every 3 weeks. Chidamide:Take 30 mg (6 tablets) each time, and take the medication twice a week, with at least 3 days between doses
  Interventions: Drug: Toripalimab; Drug: chidamide

INTERVENTIONS:
Drug: Toripalimab — Intravenous infusion, 240mg, administered once every 3 weeks, until the subject has been treated for 2 years, disease progression occurs, intolerable toxic reactions are experienced, or treatment is discontinued for other reasons.
Drug: chidamide — Take 30 mg (6 tablets) each time, and take the medication twice a week, with at least 3 days between doses (such as on Monday and Thursday, Tuesday and Friday, Wednesday and Saturday, etc.), to be taken 30 minutes after meals.

SUMMARY:
To evaluate the efficacy of Toripalimab combined with Chidamide in the treatment of relapsed/refractory peripheral T-cell lymphoma.

DETAILED DESCRIPTION:
The study is an open-label, single-arm, single-center, Phase II clinical trial. The trial design adopts the Simon optimal two-stage design. The number of effective cases in the first stage is 15; if fewer than 5 effective cases are observed, the trial will be terminated, otherwise, the trial will continue. The total sample size for the trial is at least 43 cases. All subjects receive treatment with the Toripalimab and Chidamide regimen until the subject has been treated for 2 years, disease progression occurs, intolerable toxic reactions occur, or treatment is terminated for other reasons, whichever comes first. After the end of treatment, subjects are required to complete the end-of-treatment visit within 7 days. Safety follow-up after the last dose is required at 30 days (±7 days) and 90 days (±7 days) after the last dose, with adverse event (AE) collection up to 90 days after the last dose. After the end of dosing, subjects enter the follow-up period with a telephone follow-up every 12 weeks (±7 days) to collect survival information and subsequent anti-tumor treatments until death or loss to follow-up. If a subject discontinues treatment for reasons other than PD (progressive disease), efficacy evaluation should continue at the same frequency as during the dosing period until the subject experiences PD, starts a new anti-tumor treatment, dies, or is lost to follow-up.

Treatment should be continued as long as clinical benefit is observed, until the patient is no longer tolerating it, for a maximum of 2 years of treatment. Atypical responses may be observed (for example, a temporary increase in tumor size or the appearance of new small lesions within the first few months, followed by a reduction in tumor size). If the patient's clinical symptoms are stable or continue to improve, even with preliminary evidence of disease progression, based on the overall judgment of clinical benefit, it may be considered to continue treatment with this regimen until disease progression is confirmed.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older, both males and females are eligible;
2. Histologically confirmed peripheral T-cell lymphoma (PTCL) that has relapsed or is refractory after at least one line of systemic therapy. The definitions are as follows:

   Relapse: Patients who achieved a Complete Response (CR) in previous treatments and have new lesions at the original site or elsewhere; Refractory: Patients who did not achieve CR after adequate treatment. For nasal-type NK/T-cell lymphoma, previous treatments must have included a chemotherapy regimen containing asparaginase;
3. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 2;
4. Expected survival of at least 3 months;
5. At least one measurable lesion in two dimensions, with the following criteria:

   For intra-nodular lesions: Longest diameter >1.5 cm, shortest diameter >1.0 cm; For extra-nodular lesions: Longest diameter >1.0 cm;
6. Adequate organ function as follows (no use of blood components or cytokines within 14 days before the first administration of the study drug): Hematology: Neutrophil count (NEUT) ≥ 1.5 × 10^9/L, Platelet count (PLT) ≥ 75

   * 10^9/L, Hemoglobin (HGB) ≥ 90 g/L; Liver function: Total serum bilirubin (TBIL) ≤ 1.5 × Upper Limit of Normal (ULN); Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) ≤ 2.5 × ULN; if there is liver metastasis, TBIL ≤ 3 × ULN, ALT and AST ≤ 5 × ULN; Renal function: Serum creatinine (Cr) ≤ 1.5 × ULN; Thyroid function: Thyroid-stimulating hormone (TSH) within the normal range; if TSH is abnormal, Free Triiodothyronine (FT3) and Free Thyroxine (FT4) should be within the normal range or abnormal without clinical significance;
7. Signed an informed consent form and is able to comply with the visits and procedures specified in the protocol.

Exclusion Criteria:

1. Diagnosed with Adult T-cell Leukemia/Lymphoma (ATLL);
2. Confirmed central nervous system (CNS) infiltration of lymphoma, including brain parenchymal invasion, meningeal involvement, or spinal cord compression;
3. T-cell lymphoma primarily starting extranodally in the skin, such as: Mycosis Fungoides/Sezary Syndrome (MF/SS), primary cutaneous CD30-positive T-cell lymphoproliferative disorders, primary cutaneous δγT-cell lymphoma, primary cutaneous CD8-positive aggressive, epidermotropic cytotoxic T-cell lymphoma, primary cutaneous acral CD8-positive T-cell lymphoma, lymphomatoid papulosis, primary cutaneous CD4-positive small to medium T-cell lymphoproliferative disorders;
4. Patients who have previously used PD-1 monoclonal antibodies/PD-L1 monoclonal antibodies or Chidamide;
5. Patients with certain specific past medical histories, such as active autoimmune diseases, type 1 diabetes, thyroid hormone replacement required for hypothyroidism (except Hashimoto's thyroiditis), severe mental illness;
6. Patients who require the use of immunosuppressants or systemic or absorbable local hormone therapy for immunosuppressive purposes (dose >10mg/d prednisone or other equivalent efficacy hormones) within 14 days before the first administration or during the study;
7. Patients who have received radiotherapy, chemotherapy, hormone therapy, surgery, targeted therapy, or systemic treatment with antibody drugs within 4 weeks before the first administration; those who have used monoclonal antibody conjugated with radioactive isotopes or cytotoxins within 10 weeks before the first administration; patients who have not recovered to ≤grade 1 toxicity from previous anti-tumor treatments (except for alopecia);
8. Patients with uncontrolled hypertension (systolic blood pressure ≥180mmHg and/or diastolic blood pressure ≥100mmHg);
9. Patients who have undergone autologous stem cell transplantation within 3 months before the first administration;
10. Patients with a history of organ transplantation or allogeneic bone marrow transplantation;
11. Patients who have received or plan to receive live attenuated vaccines within 4 weeks before the first administration or during the study;
12. Patients with a history of allergy to macromolecular protein preparations or anti-PD-1 antibodies;
13. Patients with a history of or concurrent other malignant tumors (except for skin basal cell carcinoma and cervical carcinoma in situ that have been cured for more than 3 years);
14. Patients with uncontrollable or severe cardiovascular diseases, those who have had New York Heart Association (NYHA) class II or above congestive heart failure, unstable angina, myocardial infarction, and other cardiovascular diseases within 6 months before the first administration;
15. HIV-positive patients, or those with active hepatitis (for hepatitis B: reference to hepatitis B five items and HBV-DNA, transaminases, etc., for hepatitis C: reference to HCV antibodies and HCV RNA);
16. Patients who have received any other clinical trial drugs/devices within 4 weeks before the first administration;
17. Patients with a history of drug abuse or alcoholism within 6 months before the first administration;
18. Patients with a history of or concurrent interstitial lung disease (except for interstitial lung disease caused by radiochemotherapy and currently asymptomatic);
19. Patients with active infections requiring systemic treatment;
20. Patients with active pulmonary tuberculosis infection;
21. Pregnant or lactating women;
22. Patients deemed unsuitable for enrollment by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2024-04-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 24months
  The primary efficacy endpoint will be assessed based on the Lugano 2014 criteria for Objective Response Rate (ORR), which includes both Complete Response (CR) and Partial Response (PR).

SECONDARY OUTCOMES:
Overall Survival (OS) | 24months
  The time from the start of the trial to death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medical Oncology, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided